CLINICAL TRIAL: NCT03319485
Title: A Pivotal Clinical Trial of the Management of the Medically-Refractory Dyskinesia Symptoms or Motor Fluctuations of Advanced Idiopathic Parkinson's Disease With Unilateral Lesioning of the Globus Pallidum Using the ExAblate Neuro System
Brief Title: ExAblate Pallidotomy for Medically-Refractory Dyskinesia Symptoms or Motor Fluctuations of Advanced Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PD006
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: ExAblate; MRgFUS; Pallidotomy
MeSH Terms: conditions — Parkinson Disease | interventions — Pallidotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ExAblate Pallidotomy (Experimental): ExAblate treatment for Advanced Idiopathic Parkinson's Disease
  Interventions: Device: ExAblate Pallidotomy
- Sham ExAblate Pallidotomy (Sham Comparator): Sham (fake) treatment
  Interventions: Device: Sham ExAblate Pallidotomy

INTERVENTIONS:
Device: ExAblate Pallidotomy — ExAblate Pallidotomy for Parkinson's Disease
  Other Names: MRgFUS; Pallidotomy
  Arms: ExAblate Pallidotomy
Device: Sham ExAblate Pallidotomy — ExAblate MRgFUS Sham Procedure
  Arms: Sham ExAblate Pallidotomy

SUMMARY:
Evaluate the safety and efficacy of unilateral focused ultrasound pallidotomy using the ExAblate 4000 System in the management of dyskinesia symptoms or motor fluctuations for medication refractory, advanced idiopathic Parkinson's disease.

DETAILED DESCRIPTION:
The goal of this prospective, two-arm, sham-controlled, randomized, multi-center pivotal study is to evaluate the safety and efficacy of unilateral focused ultrasound pallidotomy using the ExAblate 4000 System in the management of dyskinesia symptoms or motor fluctuations for medication refractory, advanced idiopathic Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 30 years and older.
2. Subjects who are able and willing to give informed consent and able to attend all study visits through 12 Months.
3. Subjects with a diagnosis of idiopathic PD by UK Brain Bank Criteria as confirmed by a movement disorder neurologist at the site.
4. Levodopa responsive as defined by at least a 30% reduction in MDS-UPDRS motor subscale in the ON vs OFF medication state.
5. MDS-UPDRS score of ≥ 20 in the meds OFF condition OR Motor complications of PD on optimum medical treatment .
6. Subjects should be on a stable dose of all PD medications for 30 days prior to study entry as determined by medical records.
7. Subject is able to communicate sensations during the ExAblate procedure.
8. Subjects on stable antidepressant medications for at least 3 months

Exclusion Criteria:

1. Hoehn and Yahr stage in the ON medication state of 3 or greater.
2. Presence of other central neurodegenerative disease suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease.
3. Any suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications.
4. Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia.
5. Presence of significant cognitive impairment using MMSE ≤ 24.
6. Unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation.
7. Subjects with an active alcohol or drug dependency or history of drug/alcohol abuse within the past year
8. Subjects with unstable cardiac status
9. Severe hypertension (diastolic BP > 100 on medication).
10. Current medical condition resulting in abnormal bleeding and/or coagulopathy.
11. Receiving anticoagulant (e.g., warfarin) or antiplatelet (e.g., aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g., Avastin) within one month of focused ultrasound procedure.
12. Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter; a documented clinical coagulopathy; or INR coagulation studies exceeding the institution's laboratory standard
13. Patient with kidney disease or on dialysis.
14. Subjects with standard contraindications for MR imaging
15. Significant claustrophobia that cannot be managed with mild medication.
16. Subjects who weigh more than the upper weight limit of the MR scanner table and who cannot fit into the MR scanner.
17. Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment.
18. History of intracranial hemorrhage, multiple strokes, or a stroke within past 6 months.
19. Subjects with a history of seizures within the past year.
20. Subjects with brain tumors.
21. Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment.
22. Are participating or have participated in another clinical trial in the last 30 days.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Responder Analysis | Change in UDysRS and MDS-UPDRS Part III Motor Exam score from before treatment to 3 months following treatment
  Responder is defined as the patient reaching a minimally clinically significant difference on: 1. UDysRS (this measures dyskinesia and their impact) OR 2. MDS-UPDRS Part III Motor Exam -Total score (this measures overall motor fluctuations).

SECONDARY OUTCOMES:
Severity of Device and Procedure related complications | At the time of ExAblate Pallidotomy procedure
  To evaluate of the incidence and severity of device- and procedure-related

CONTACTS AND LOCATIONS:
Locations (20):
- United States (11):
  - Stanford University Medical Center, Stanford, California
  - Palm Beach Neuroscience Institute/Sperling Medical Group, Boynton Beach, Florida
  - University of Maryland Medical System, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - New York University Health Langone, New York, New York
  - Weill Cornell Medicine, New York, New York
  - The Ohio State Wexner Medical Center, Columbus, Ohio
  - Pennsylvania Hospital Department of Neurosurgery, Philadelphia, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington
- Toronto Western Hospital, Toronto, Ontario, Canada
- Rambam Health Care, Haifa, Israel
- Italy (2):
  - Fondazione IRCCS Neurological Institute Carlo Besta, Milan
  - Azienda Ospedaliera Universitaria di Verona, Univerista di Verona, Verona
- Severance Hospital, Yonsei University Health System, Seoul, South Korea
- Spain (2):
  - CINAC-Hospital HM Puerta del Sur, Móstoles, Madrid
  - Clinica Universidad De Navarra, Pamplona, Navarre
- Chang Bing Show Chwan Memorial Hospital, Changhua, Taiwan
- St. Mary's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Krishna V, Fishman PS, Eisenberg HM, Kaplitt M, Baltuch G, Chang JW, Chang WC, Martinez Fernandez R, Del Alamo M, Halpern CH, Ghanouni P, Eleopra R, Cosgrove R, Guridi J, Gwinn R, Khemani P, Lozano AM, McDannold N, Fasano A, Constantinescu M, Schlesinger I, Dalvi A, Elias WJ. Trial of Globus Pallidus Focused Ultrasound Ablation in Parkinson's Disease. N Engl J Med. 2023 Feb 23;388(8):683-693. doi: 10.1056/NEJMoa2202721. PMID 36812432